CLINICAL TRIAL: NCT07213518
Title: High Velocity Nasal Insufflation Versus Continuous Positive Airway Pressure in COVID 19 Pneumonic Patients With Acute Type 1 Respiratory Failure
Brief Title: High Velocity Nasal Insufflation Versus Continuous Positive Airway Pressure in COVID 19 Pneumonic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS.21.08.1614
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: COVID-19 Pneumonia
Keywords: High Velocity Nasal Insufflation; Acute Type 1 Respiratory Failure; COVID 19 Pneumonic Patients; Continuous Positive Airway Pressure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Positive Airway Pressure (Active Comparator): COVID 19 Pneumonic Patients with Acute Type 1 Respiratory Failure received Continuous Positive Airway Pressure
  Interventions: Device: Continuous Positive Airway Pressure
- High Velocity Nasal Insufflation (Active Comparator): COVID 19 Pneumonic Patients with Acute Type 1 Respiratory Failure received High Velocity Nasal Insufflation
  Interventions: Device: High Velocity Nasal Insufflation

INTERVENTIONS:
Device: High Velocity Nasal Insufflation — COVID 19 Pneumonic Patients with Acute Type 1 Respiratory Failure received High Velocity Nasal Insufflation
  Arms: High Velocity Nasal Insufflation
Device: Continuous Positive Airway Pressure — COVID 19 Pneumonic Patients with Acute Type 1 Respiratory Failure received Continuous Positive Airway Pressure
  Arms: Continuous Positive Airway Pressure

SUMMARY:
compare the efficacy of High-Velocity Nasal Insufflation (HVNI) versus Continuous Positive Airway Pressure (CPAP) in managing COVID 19 pneumonic patients with acute type 1 respiratory failure

DETAILED DESCRIPTION:
A prospective randomized controlled trial was conducted on 108 patients with COVID 19 pneumonia with acute hypoxemic respiratory failure at Mansoura University Hospitals to compare the efficacy of High-Velocity Nasal Insufflation (HVNI) versus Continuous Positive Airway Pressure (CPAP) in managing COVID 19 pneumonic patients with acute type 1 respiratory failure, focusing on the need for invasive mechanical ventilation (IMV) and 28-day mortality. Patients were randomized into two equal groups: HVNI group and CPAP group. Baseline characteristics, respiratory parameters, and clinical outcomes were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years with COVID 19 pneumonia with acute type 1 respiratory failure were included.

Exclusion Criteria:

* patients with hypercapnic respiratory failure.
* patients with a disturbed level of consciousness and/or a high risk of aspiration
* individuals with hypotension
* patients requiring invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Correction of hypoxia in COVID 19 Pneumonic Patients with Acute Type 1 Respiratory Failure | 6 months
  assessment of efficacy of High Velocity Nasal Insufflation versus Continuous Positive Airway Pressure in COVID 19 Pneumonic Patients with Acute Type 1 Respiratory Failure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt